CLINICAL TRIAL: NCT04764058
Title: Efficacy and Safety of Colistin Based Antibiotic Therapy for Multidrug Resistant Gram Negative Infections in Pediatric Intensive Care Unit
Brief Title: Efficacy and Safety of Colistin Based Antibiotic Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Saeed Attia Mancy, Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 210
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Septicemia; Bacterial Infections
MeSH Terms: conditions — Sepsis; Bacterial Infections | interventions — Cilastatin, Imipenem Drug Combination; Meropenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montherapy (Other): Thirty patients will receive IV Imipenem in doses of 15 to 25 mg/kg every 6 hours
  Interventions: Drug: Tienam 500; Device: Infusion
- Combination (Other): Thirty patients will receive IV Colistin in dosages of 50,000-75,000 IU/kg/day in three divided doses, infused IV in 10mL normal saline over 30 minutes with IV Imipenem in doses of 15 to 25 mg/kg every 6 hours¬.21,22,24 Colistin formulation consists of 2 million IU per vial.
  Interventions: Drug: Tienam 500; Device: Infusion

INTERVENTIONS:
Drug: Tienam 500 — Imipenem and cilastatin sodium
  Other Names: Meronem
Device: Infusion — Health caregivers give the drug to the patients and monitoring the infusion rate

SUMMARY:
To evaluate the efficacy and safety of antibiotic combinations containing Colistin in the treatment of children with multidrug-resistant gram negative infections admitted in the pediatric surgery intensive care unit.

The main outcome measure is clinical and microbiological responses to therapy.

The secondary outcome is the occurrence of adverse events during Colistin combination treatment.

DETAILED DESCRIPTION:
Patients and Methods

Design of the study:

- Prospective, Randomized, interventional study.

Setting:

- The study will be conducted in the pediatric surgery intensive care unit in Children's Hospitals, Ain Shams University, Cairo, Egypt.

Subjects:

- Pediatric patients admitted in pediatric surgery intensive care unit.

Inclusion criteria:

All children with culture-proven nosocomial infections due to multidrug resistance gram-negative organisms

Exclusion criteria:

1. Patients who started on Colistin treatment outside the pediatric surgery intensive care unit and transferred to the unit afterward will be excluded.
2. Patients who will receive <6 doses of intravenous Colistin will be excluded.
3. Patients received Imipenem or Colistin-Imipenem compination as empirical antibiotic.

Methodology:

- Sixty pediatric patients admitted to the pediatric surgery intensive care unit will be enrolled in the study and will be randomly assigned to either Group I or Group II

Group I: Thirty patients will receive IV Colistin in dosages of 50,000-75,000 IU/kg/day in three divided doses, infused IV in 10mL normal saline over 30 minutes with IV Imipenem in doses of 15 to 25 mg/kg every 6 hours¬.21,22,24 Colistin formulation consists of 2 million IU per vial. Group II: Thirty patients will receive IV Imipenem in doses of 15 to 25 mg/kg every 6 hours¬. 22,24

For all patients the following data will be collected:

1. Demographic data (age, gender, weight).
2. The risk factors for nosocomial infections.
3. Pediatric surgery intensive care unit stay.
4. Type of surgeries performed.
5. Site of isolation of organisms.
6. The dose and duration of therapy.
7. Serum creatinine levels will be assessed at baseline, once weekly and at the end of Colistin combination therapy.
8. Nephrotoxic co-medication monitoring.
9. Clinical (resolution of signs and symptoms of infection) and
10. microbiological (bacteriologic responses) outcomes will be evaluated during treatment and at the end of the treatment.

According to the inclusion and exclusion criteria, the demographic data for the intended ICU patients was collected, then the sample was withdrawn from the infected site to be cultured on specific culture media (such as blood agar, MacConkey agar, Chocolate agar), and identification of the isolated microorganism was detected by biochemical tests and Vitek-2 compact system whenever required. Antimicrobial sensitivity to Colistin was tested using the micro broth dilution method, in order to be evaluated in Colistin therapy. After culture-proven, the drug was given, either IV Colistin-Imipenem/Cilastatin as a combination or Imipenem/Cilastatin as a monotherapy. Throughout this step, the hemodynamic parameters were measured during the process of treatment, without neglecting the serum creatinine level to detect any nephrotoxicity.

We assure the right drug handling, dosing, dispensing, and monitoring. At the end of the treatment, the duration and length of PICU stay were recorded.

The decision and/or conclusion of treatment failure and/ or success was based upon the worsening and/or improvement of the patients' parameters and their situation including the results of the microbiological examination before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* All children with culture proven nosocomial infections due to multidrug resistance gram-negative organisms

Exclusion Criteria:

* 1. Patients who started on Colistin treatment outside the pediatric surgery intensive care unit and transferred to the unit afterward will be excluded.

  2. Patients who will receive <6 doses of intravenous Colistin will be excluded.

  3. Patients received Imipenem or Colistin-Imipenem compination as empirical antibiotic.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Parameters Measurement ,heart beating rate. | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the heart beating rate.
Hemodynamic Parameters Measurement ,body temperature | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the body temperature
Hemodynamic Parameters Measurement ,respiratory rate. | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the respiratory rate.
Hemodynamic Parameters Measurement ,blood pressure | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the blood pressure
Hemodynamic Parameters Measurement ,partial oxygen saturation pressure | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the partial oxygen saturation pressure
Hemodynamic Parameters Measurement and Septic Markers, serum lactate | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the serum lactate
Hemodynamic Parameters Measurement ,serum creatinine | 2 year
  the efficacy and safety of antibiotic combination containing Colistin. We will monitor the serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: AHMED S ATTIA, Principal Investigator — Heliopolis University
Locations (1):
- Ain Shams Univesity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No